CLINICAL TRIAL: NCT03306251
Title: ANRS CO11 : National Cohort of Children Born to HIV-positive Mothers
Brief Title: National Cohort of Children Born to HIV-positive Mothers
Acronym: EPF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS-CO11-EPF
Record Dates: First submitted 2016-09-20; First posted 2017-10-11 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Mother to Child Transmission of HIV
Keywords: HIV; Pregnancy; Prevention of mother-to-child transmission

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to provide a surveillance system to monitor changes in the rate of mother to child HIV transmission and preventive practices in France and especially to identify the occurrence of toxicity in children exposed perinatally to antiretroviral drugs.

DETAILED DESCRIPTION:
The goal of the CO11 national cohort is to provide with CO1 a wider surveillance system to monitor changes in the rate of mother to child transmission and preventive practices in France and especially to identify the occurrence of toxicity in children exposed perinatally to antiretroviral drugs.

The CO11 EPF enrolle HIV infected women who delivery in maternity generally smaller than CO1 maternity (15 sites in Paris area, 35 in mainland France and 4 in the DOM).

Maternal clinical, biological and therapeutic data before and during pregnancy were collected at delivery, with simplified questionnaires.

The children are examined clinically and biologically at birth, 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women >= 18 years
* infected with HIV1 and/or HIV2

Exclusion Criteria:

* guardianship or judicial or administrative detention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion as soon as possible during pregnancy of HIV-women in obstetrical sites (15 sites in Paris area, 35 in mainland France and 4 in the DOM)
Sampling Method: Non-Probability Sample
Enrollment: 5200 (Estimated)
Dates: Start 2005-06; Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PMTCT strategies by measuring rate of mother to child transmission of HIV | At birth up to 24 months
  Number of infected children (HIV RNA >50c/mL or Positive serology) reported on the total number of children

SECONDARY OUTCOMES:
Immuno-virological response during pregnancy | At inclusion up to childbirth
  HIV ARN <50c/mL, CD4 cells count>500 cells/mL
Tolerance and toxicity of different kind of MTCT prophylaxis during pregnancy | At inclusion up to childbirth
  incidence of pathologies during pregnancy
Impact of different kind of MTCT prophylaxis on childbirth | At delivery
  Childbirth mode (Number of emergency Caesarean section, Number of planned caesarean section)
Impact of different kind of MTCT prophylaxis during pregnancy on uninfected children | At childbirth, 1 month, 3 months, 6 months, 12 months and 18-24 months
  Clinical abnormalities (occurrence of adverse events)

CONTACTS AND LOCATIONS:
Overall Officials: Josiane WARSZAWSKI, Principal Investigator — CESP INSERM U1018
Locations (52):
- France (49):
  - CHU Hôpital Nord, Amiens
  - Centre Hospitalier Universitaire, Angers
  - Centre Hosipitalier, Annecy
  - Centre Hospitalier Robert Ballanger, Aulnay
  - Centre Hospitalier Général de Bastia, Bastia
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHRU Saint Jacques, Besançon
  - Centre hospitalier de Béziers, Béziers
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Centre Hospitalier Régional Universitaire de Brest, Brest
  - CHRU Clemenceau, Caen
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre Hospitalier Général, Creil
  - CHRU de Dijon, Dijon
  - Centre Hospitalier Général, Évreux
  - Centre Hospitalier Général, Fontainebleau
  - Centre Hospitalier Les Oudayries, La Roche-sur-Yon
  - Centre Hospitalier de Lagny, Lagny-sur-Marne
  - Hôpital André Mignot, Versailles, Le Chesnay
  - Centre Hospitalier Universitaire, Limoges
  - Centre Hospitalier Général, Longjumeau
  - Centre Hospitalier Bretagne Sud, Lorient
  - Centre Hospitalier François Quesnay, Mantes-la-Jolie
  - Centre Hospitalier de Meaux, Maux
  - Centre Hospitalier Marc Jacquet, Melun
  - Centre Hospitalier Intercommunal, Montfermeil
  - CHU Nancy, Nancy
  - CHU Caremeau, Nîmes
  - Centre Hospitalier Régional, Orléans
  - Centre Hospitalier Général, Orsay
  - Bon secours-Saint Joseph, Paris
  - CHG Maréchal Joffre, Perpignan
  - Centre Hospitalier Intercommunal, Poissy
  - Centre Hospitalier René Dubos, Pontoise
  - Centre Hospitalier Léon Binet, Provins
  - Hôpital Laennec, Quimper
  - CHR American Memorial Hospital, Reims
  - CHU Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Centre Hopsitalier Yves Le Foll, Saint-Brieuc
  - Hôpital Bellevue, Saint-Etienne
  - Centre hospitalier, Saint-Julien
  - Hôpital de Saint-Martin, Saint-Martin
  - Centre Hospitalier de Saint Nazaire-Cité Sanitaire, Saint-Nazaire
  - Hôpital Font Pré, Toulon
  - CHRU de Tours, Tours
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Centre Hospitalier, Vernon
  - Centre Hospitalier Intercommunal, Villeneuve-Saint-Georges
- CHG de Cayenne, Cayenne, French Guiana
- CHU Pointe à Pitre, Les Abymes, Pointe-à-Pitre, Guadeloupe
- Hôpital Victor Fouche, Fort-de-France, Martinique

REFERENCES:
- [Result] Mandelbrot L, Tubiana R, Le Chenadec J, Dollfus C, Faye A, Pannier E, Matheron S, Khuong MA, Garrait V, Reliquet V, Devidas A, Berrebi A, Allisy C, Elleau C, Arvieux C, Rouzioux C, Warszawski J, Blanche S; ANRS-EPF Study Group. No perinatal HIV-1 transmission from women with effective antiretroviral therapy starting before conception. Clin Infect Dis. 2015 Dec 1;61(11):1715-25. doi: 10.1093/cid/civ578. Epub 2015 Jul 21. PMID 26197844
- [Result] Taron-Brocard C, Le Chenadec J, Faye A, Dollfus C, Goetghebuer T, Gajdos V, Labaune JM, Perilhou A, Mandelbrot L, Blanche S, Warszawski J; France REcherche Nord&Sud Sida-HIV Hepatites - Enquete Perinatale Francaise - CO1/CO11 Study Group. Increased risk of serious bacterial infections due to maternal immunosuppression in HIV-exposed uninfected infants in a European country. Clin Infect Dis. 2014 Nov 1;59(9):1332-45. doi: 10.1093/cid/ciu586. Epub 2014 Jul 22. PMID 25053719
- [Result] Sibiude J, Mandelbrot L, Blanche S, Le Chenadec J, Boullag-Bonnet N, Faye A, Dollfus C, Tubiana R, Bonnet D, Lelong N, Khoshnood B, Warszawski J. Association between prenatal exposure to antiretroviral therapy and birth defects: an analysis of the French perinatal cohort study (ANRS CO1/CO11). PLoS Med. 2014 Apr 29;11(4):e1001635. doi: 10.1371/journal.pmed.1001635. eCollection 2014 Apr. PMID 24781315
- [Result] Briand N, Jasseron C, Sibiude J, Azria E, Pollet J, Hammou Y, Warszawski J, Mandelbrot L. Cesarean section for HIV-infected women in the combination antiretroviral therapies era, 2000-2010. Am J Obstet Gynecol. 2013 Oct;209(4):335.e1-335.e12. doi: 10.1016/j.ajog.2013.06.021. Epub 2013 Jun 18. PMID 23791563
- [Result] Briand N, Warszawski J, Mandelbrot L, Dollfus C, Pannier E, Cravello L, Nguyen R, Matheron I, Winer N, Tubiana R, Rouzioux C, Faye A, Blanche S; ANRS-EPF CO1-CO11 Study Group. Is intrapartum intravenous zidovudine for prevention of mother-to-child HIV-1 transmission still useful in the combination antiretroviral therapy era? Clin Infect Dis. 2013 Sep;57(6):903-14. doi: 10.1093/cid/cit374. Epub 2013 May 31. PMID 23728147
- [Result] Rachas A, Warszawski J, Le Chenadec J, Legeai C, Teglas JP, Goujard C, Rouzioux C, Mandelbrot L, Tubiana R, Meyer L. Does pregnancy affect the early response to cART? AIDS. 2013 Jan 28;27(3):357-67. doi: 10.1097/QAD.0b013e32835ac8bc. PMID 23079802
- [Result] Jasseron C, Mandelbrot L, Dollfus C, Trocme N, Tubiana R, Teglas JP, Faye A, Rouzioux C, Blanche S, Warszawski J. Non-disclosure of a pregnant woman's HIV status to her partner is associated with non-optimal prevention of mother-to-child transmission. AIDS Behav. 2013 Feb;17(2):488-97. doi: 10.1007/s10461-011-0084-y. PMID 22130651
- [Result] Simon A, Warszawski J, Kariyawasam D, Le Chenadec J, Benhammou V, Czernichow P, Foissac F, Laborde K, Treluyer JM, Firtion G, Layouni I, Munzer M, Bavoux F, Polak M, Blanche S; ANRS French Perinatal Cohort Study Group. Association of prenatal and postnatal exposure to lopinavir-ritonavir and adrenal dysfunction among uninfected infants of HIV-infected mothers. JAMA. 2011 Jul 6;306(1):70-8. doi: 10.1001/jama.2011.915. PMID 21730243
- [Result] Sibiude J, Warszawski J, Tubiana R, Dollfus C, Faye A, Rouzioux C, Teglas JP, Ekoukou D, Blanche S, Mandelbrot L. Premature delivery in HIV-infected women starting protease inhibitor therapy during pregnancy: role of the ritonavir boost? Clin Infect Dis. 2012 May;54(9):1348-60. doi: 10.1093/cid/cis198. Epub 2012 Mar 28. PMID 22460969
- [Result] Tubiana R, Le Chenadec J, Rouzioux C, Mandelbrot L, Hamrene K, Dollfus C, Faye A, Delaugerre C, Blanche S, Warszawski J. Factors associated with mother-to-child transmission of HIV-1 despite a maternal viral load <500 copies/ml at delivery: a case-control study nested in the French perinatal cohort (EPF-ANRS CO1). Clin Infect Dis. 2010 Feb 15;50(4):585-96. doi: 10.1086/650005. PMID 20070234
- [Result] Briand N, Mandelbrot L, Le Chenadec J, Tubiana R, Teglas JP, Faye A, Dollfus C, Rouzioux C, Blanche S, Warszawski J; ANRS French Perinatal Cohort. No relation between in-utero exposure to HAART and intrauterine growth retardation. AIDS. 2009 Jun 19;23(10):1235-43. doi: 10.1097/QAD.0b013e32832be0df. PMID 19424054
- [Result] Mandelbrot L, Jasseron C, Ekoukou D, Batallan A, Bongain A, Pannier E, Blanche S, Tubiana R, Rouzioux C, Warszawski J; ANRS French Perinatal Cohort (EPF). Amniocentesis and mother-to-child human immunodeficiency virus transmission in the Agence Nationale de Recherches sur le SIDA et les Hepatites Virales French Perinatal Cohort. Am J Obstet Gynecol. 2009 Feb;200(2):160.e1-9. doi: 10.1016/j.ajog.2008.08.049. Epub 2008 Nov 4. PMID 18986640
- [Result] Jasseron C, Mandelbrot L, Tubiana R, Teglas JP, Faye A, Dollfus C, Le Chenadec J, Rouzioux C, Blanche S, Warszawski J; ANRS French Perinatal Cohort. Prevention of mother-to-child HIV transmission: similar access for sub-Sahara African immigrants and for French women? AIDS. 2008 Jul 31;22(12):1503-11. doi: 10.1097/QAD.0b013e3283065b8c. PMID 18614874
- [Result] Benhammou V, Warszawski J, Bellec S, Doz F, Andre N, Lacour B, Levine M, Bavoux F, Tubiana R, Mandelbrot L, Clavel J, Blanche S; ANRS-Enquete Perinatale Francaise. Incidence of cancer in children perinatally exposed to nucleoside reverse transcriptase inhibitors. AIDS. 2008 Oct 18;22(16):2165-77. doi: 10.1097/QAD.0b013e328311d18b. PMID 18832880
- [Result] Warszawski J, Tubiana R, Le Chenadec J, Blanche S, Teglas JP, Dollfus C, Faye A, Burgard M, Rouzioux C, Mandelbrot L; ANRS French Perinatal Cohort. Mother-to-child HIV transmission despite antiretroviral therapy in the ANRS French Perinatal Cohort. AIDS. 2008 Jan 11;22(2):289-99. doi: 10.1097/QAD.0b013e3282f3d63c. PMID 18097232